CLINICAL TRIAL: NCT03566550
Title: A Case-Control, Observational Study of the Postprandial Changes in Magnetic Resonance Imaging Parameters of Gastrointestinal Function and Transit in People With Cystic Fibrosis
Brief Title: Gut Imaging for Function & Transit in Cystic Fibrosis Study 1
Acronym: GIFT-CF1
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18GA006
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Results first posted 2021-04-05 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CF: people with cystic fibrosis
  Interventions: Diagnostic Test: MRI scans
- Control: people without cystic fibrosis
  Interventions: Diagnostic Test: MRI scans

INTERVENTIONS:
Diagnostic Test: MRI scans — Repeated MRI scans imaging digestion of standard meals

SUMMARY:
Many people with Cystic Fibrosis (CF) are troubled by symptoms from their stomach and bowels: their gastrointestinal (GI) tract. Symptoms affect quality of life and can also reduce people's ability to digest enough calories to remain healthy, leaving them undernourished and less able to deal with other health problems such as infection.

Clinical tests to assess bowel function are limited. Many tests involve inserting a sensor or camera into the bowel, so they are not suitable for long periods, and can be uncomfortable. In Nottingham the investigators have developed imaging scans which can assess how someone's digestion works without any invasive device. The type of scanning the investigators use is called Magnetic Resonance Imaging, or MRI.

The purpose of this study is to see if those scanning methods can be used in people with CF to understand their digestion and any problems they have.

DETAILED DESCRIPTION:
This is a small pilot study to establish that differences in digestion between people with and without CF can be quantified by repeated MR scans in fasted participants in response to standardised meals.

Participants will complete questionnaires on gastrointestinal function and symptoms: the PAC-SYM questionnaire, validated to assess symptom burden in adults with chronic constipation; and the CF abdomen questionnaire, developed in German for use in young people and adults with cystic fibrosis.

After this, participants only need to attend one study day at the Sir Peter Mansfield Imaging Centre. On this day they will be asked to withhold any medicines specifically targeted to alter bowel habit. This shall include laxatives but not enzyme replacement therapy. They should attend on the study day having fasted since waking, other than water for essential medicines.

They will have their first MRI scan fasted. After the scan they will eat a standard test meal, and be scanned again first at half hour, then hour intervals until six hours after the first meal. The final scan will constitute the end of the study for each participant. Each session in the MRI scanner will last around 15 minutes. After each scan they will complete a validated rating scale for any current symptoms: the Gastrointestinal Symptom Rating Scale (GSRS).In between scans, participants will have access to a lounge with wifi and a television.

Infection control requirements mean that the investigators are unable to scan more than one patient with CF on a single day. Patient scans will alternate with those of a Control participant. The investigators will aim to frequency match Controls with Patients for age and gender.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 - 40 years
* Capacity to consent, or to understand the requirements of the study where parental consent is needed
* PATIENTS: confirmed diagnosis of Cystic Fibrosis, either by sweat test or genetic testing; to reduce heterogeneity, we will only enrol homozygous CF patients with the most common CFTR mutation, p.Phe508del
* CONTROLS: no clinical evidence or suspicion of Cystic Fibrosis

Exclusion Criteria:• Measurement of Forced Expiratory Volume in 1 second (FEV1) of <40% predicted using Global Lung Initiative criteria, according to clinical records

* Contra-indication to MRI scanning, such as embedded metal, pacemaker
* Unable to stop medications directly prescribed to alter bowel habit, such as laxatives of anti-diarrhoeals, on the study day
* Previous resection of any part of the gastro-intestinal tract apart from appendicectomy or cholecystectomy. Surgical relief of distal ileal obstruction syndrome or neonatal ileus will be permitted unless clinical records show excision of intestine >20cm in length.
* Intestinal stoma
* Diagnosis of inflammatory bowel disease or coeliac disease confirmed by biopsy
* Gastrointestinal malignancy
* Unable to comply with dietary restrictions required for the study

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Nottingham and surrounding towns
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Smyth, Prof, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals National Health Service Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data outside the research team at this time.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 CF patients were eligible. CF patients were approached in order of their hospital attendance and the first 12 to provide written consent were enroled into the study. 13 declined to participate and 2 withdrew consent as they did not like the standardised meals or MRI.
  12 CF patients and 12 controls completed the protocol without any adverse events. 1 further control was withdrawn and replaced as the participant was unable to complete the first standardised meal and the remaining 10 MRI scans.
Groups:
- Cystic Fibrosis: people with cystic fibrosis
  MRI scans: Repeated MRI scans imaging digestion of standard meals
Period: Overall Study
Arm/Group | Cystic Fibrosis | Control
Started | 12 | 13
Completed | 12 | 12
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cystic Fibrosis | Control | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 5 | 10
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12 | 12 | 24
Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 56 [53 to 59] | 62 [59 to 75] | 59 [54 to 63]
Height (cm) [Median (Inter-Quartile Range); unit: cm] | 166 [158 to 175] | 166 [160 to 176] | 166 [158 to 176]

OUTCOME MEASURES:

1. Primary Outcome: Orocaecal Transit Time
Description: time taken after eating for ingested food to be identifiable in the caecum on MRI
Time Frame: 1 day of scanning
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Cystic Fibrosis | Control
Number analyzed (Participants) | 12 | 12
minutes | 330 [270 to NA] — please note the upper quartile for the cystic fibrosis group states NA due to censored data after 360 minutes (MRI scans were only performed until 360 minutes). | 210 [173 to 315]
Statistical Analysis 1: Comparison: Cystic Fibrosis vs Control; Test type: Other; p = 0.04, Log Rank

2. Secondary Outcome: Gastric Half Emptying Times
Description: volume of stomach at each time point of digestion to measure speed of gastric emptying (time taken for half the gastric contents to be emptied)
Time Frame: 1 day of scanning
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Cystic Fibrosis | Control
Number analyzed (Participants) | 12 | 12
minutes | 97 [71 to 128] | 80 [66 to 88]
Statistical Analysis 1: Comparison: Cystic Fibrosis vs Control; Test type: Other; p = 0.3, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Small Bowel Water Content (Corrected for Body Surface Area)
Description: volume of water content in small bowel representing secretions (area under the curve - timepoints at baseline then 0,30,60,90,120,150,180,240,300,360 minutes)
Time Frame: 1 day of scanning
Measure: Median (Inter-Quartile Range); unit: L.min/m^2
Arm/Group | Cystic Fibrosis | Control
Number analyzed (Participants) | 12 | 12
L.min/m^2 | 62 [36 to 80] | 34 [28 to 41]
Statistical Analysis 1: Comparison: Cystic Fibrosis vs Control; Test type: Other; p = 0.021, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Colonic Volume (Corrected for Body Surface Area)
Description: volume of colon representing ease of chyme passage through colon (area under the curve - timepoints at baseline then 0,30,60,90,120,150,180,240,300,360 minutes)
Time Frame: 1 day of scanning
Measure: Median (Inter-Quartile Range); unit: L.min/m^2
Arm/Group | Cystic Fibrosis | Control
Number analyzed (Participants) | 12 | 12
L.min/m^2 | 186 [166 to 206] | 123 [89 to 146]
Statistical Analysis 1: Comparison: Cystic Fibrosis vs Control; Test type: Other; p = 0.012, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Gastrointestinal Symptoms
Description: gastrointestinal symptoms as measured by questionnaires to monitor relationship with outcomes measured by MRI. Scale of the CFAbd-score ranges from 0-100. A low score indicates fewer gastrointestinal symptoms whilst a higher score indicates more severe and frequent gastrointestinal symptoms.
Time Frame: 1 day of scanning
Measure: Median (Inter-Quartile Range); unit: CFAbd-Score units
Arm/Group | Cystic Fibrosis | Control
Number analyzed (Participants) | 12 | 12
CFAbd-Score units | 16 [5 to 25] | 7 [3 to 14]
Statistical Analysis 1: Comparison: Cystic Fibrosis vs Control; Test type: Other; p = 0.13, Wilcoxon (Mann-Whitney)

6. Other Pre Specified Outcome: T1 Relaxation Time of Ascending Colon Chyme
Description: An approximate measure of water content in chyme present in the ascending colon
Time Frame: 1 day of scanning
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Fat Fraction of the Ascending Colon Chyme
Description: A measure of fat content in chyme present in the ascending colon
Time Frame: 1 day of scanning
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 day of MRI scanning
Arm/Group | Cystic Fibrosis | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT03566550/Prot_SAP_000.pdf